CLINICAL TRIAL: NCT01672294
Title: Caregiver Outlook: An Intervention to Improve Caregiving in Serious Illness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IIR 11-347
Record Dates: First submitted 2012-05-11; First posted 2012-08-24 (Estimated); Results first posted 2017-04-17 (Actual); Last update posted 2017-04-17 (Actual); Status verified 2017-03

CONDITIONS: Heart Failure; Pulmonary Disease; Cancer
Keywords: caregiver; end of life; self-disclosure
MeSH Terms: conditions — Heart Failure; Lung Diseases; Neoplasms; Death

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- treatment (Experimental): three facilitator-led end-of-life preparation and completion sessions with a facilitator with both patient and caregiver
  Interventions: Other: Preparation and life completion
- attention control (Active Comparator): three facilitator led sessions of listening to a relaxation CD.
  Interventions: Other: Attention Control

INTERVENTIONS:
Other: Preparation and life completion — Caregiver subjects will discuss life review, issues of forgiveness and heritage and legacy.
  Arms: treatment
Other: Attention Control — Caregiver subjects will listen to a non-guided relaxation CD with facilitator.
  Arms: attention control

SUMMARY:
Informal caregivers provide a majority of care for patients during serious illness. Lack of preparation and completion may leave caregivers less capable of caring for a loved one or making crucial decisions influencing care.

This study will examine whether a preparation and completion intervention reduces caregiver anxiety, depression, anticipatory grief, and burden and improves patient quality of life and health care use.

DETAILED DESCRIPTION:
The investigators propose a randomized control trial to evaluate an intervention of preparation and completion with Veterans and their caregivers during serious illness. Specific aims are to 1) Evaluate the impact of the caregiver Outlook intervention on caregiver anxiety, depression, anticipatory grief, completion, and burden; 2) Evaluate the impact of the home versus in hospital, emergency department, or nursing facility; 3) Evaluate the impact of the intervention session's qualitative content, examining variation associated with selected demographic variables, quality of family communication, and stage of illness on change.

Caregivers in the first group ("Treatment", or "Preparation and life completion") will meet with a facilitator three times for a period of forty-five minutes each. In the first session, subjects will be asked to discuss issues related to relationship life review.

In session two, participants will be asked to speak in more depth about issues such as regret and forgiveness. In the final session, subjects will focus on legacy and celebration. Caregivers in the second group ("attention control" or "relaxation meditation") will meet with a facilitator three times for a period of forty-five minutes each and be asked to listen to a non-guided relaxation compact disk (CD) or participate in a guided relaxation exercise.

Participants in both groups will receive pre and post-test measures administered by a blinded interviewer. Outcome measures will be measures by the Functional Assessment of Cancer Therapy - General (FACT-G), Quality of life scale, FACIT-sp sub-scale, Anticipatory Grief Scale, Caregiver Reaction Assessment, the Qual-E completion and preparation sub-scales, and patient days at home.

ELIGIBILITY:
Inclusion Criteria:

* Patients with advanced cancer/Congestive heart failure/COPD/End stage renal disease who have a primary caregiver. Caregivers of Durham VAMC patients with advanced disease.

Exclusion Criteria:

* No caregiver present.
* Caregiver with Cognitive impairment/inability to speak on phone/non-English speaking

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 286 (Actual)
Dates: Start 2013-06; Primary Completion 2015-12 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen E Steinhauser, PhD, Principal Investigator — Durham VA Medical Center, Durham, NC
Locations (1):
- Durham VA Medical Center, Durham, NC, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study conducted recruitment from June 2013 to October 2015. Potential patients were identified by data pulls and then medical record review as well as obtaining approval to approach from providers. Patients were approached both at select outpatient clinics at the Durham VAMC as well as being sent invitation letters with subsequent phone calls.
Pre-assignment Details: Participant pairs (seriously-ill veteran and primary informal caregiver) were consented and then each completed a baseline interview before the dyad was randomized. Enrolled participants may be excluded if either of the pair refused to consent or did not complete a baseline.
Groups:
- Caregiver Outlook - Caregiver; Caregiver Outlook - Patient: Intervention: Three facilitator-led preparation and life completion sessions with caregiver. Intervention: Three facilitator-led preparation and life completion sessions with caregiver.
  Topics included life review, issues of forgiveness and heritage and legacy.
- Relaxation Meditation - Caregiver; Relaxation Meditation - Patient: Attention Control: Three facilitator led sessions of caregivers listening to a non-guided relaxation CD.
Period: Overall Study
Arm/Group | Caregiver Outlook - Caregiver | Caregiver Outlook - Patient | Relaxation Meditation - Caregiver | Relaxation Meditation - Patient
Started | 71 | 71 | 72 | 72
Completed | 65 | 50 | 61 | 59
Not Completed | 6 | 21 | 11 | 13
Not completed — Withdrawal by Subject | 4 | 4 | 4 | 4
Not completed — Excluded by study | 1 | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 16 | 7 | 9

BASELINE CHARACTERISTICS:
Groups:
- Caregiver Outlook - Caregiver; Caregiver Outlook - Patient: Intervention: Three facilitator-led preparation and life completion sessions with caregiver. Topics included life review, issues of forgiveness and heritage and legacy.
- Total: Total of all reporting groups
Arm/Group | Caregiver Outlook - Caregiver | Caregiver Outlook - Patient | Relaxation Meditation - Caregiver | Relaxation Meditation - Patient | Total
Number analyzed (Participants) | 71 | 71 | 72 | 72 | 286
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.8 (11.32) | 66.8 (7.85) | 60.1 (12.05) | 65.4 (9.21) | 63.3 (10.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67 | 4 | 67 | 3 | 141
  Male | 4 | 67 | 5 | 69 | 145
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 2 | 0 | 7
  Not Hispanic or Latino | 68 | 69 | 68 | 72 | 277
  Unknown or Not Reported | 0 | 0 | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants] — NIH/OMB categories collapsed to: African-American\Black, Caucasian\White Other including more than 1 race, missing
  Participants
    American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
    Asian | 0 | 0 | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
    Black or African American | 31 | 29 | 30 | 32 | 122
    White | 36 | 38 | 33 | 38 | 145
    More than one race | 4 | 4 | 7 | 2 | 17
    Unknown or Not Reported | 0 | 0 | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 71 | 71 | 72 | 72 | 286
Dyad Relationship [Count of Participants; unit: Participants] — Respective relationship of participant to other dyad in pair.
  Participants
    Spouse | 52 | 52 | 53 | 53 | 210
    Adult Child | 6 | 2 | 3 | 1 | 12
    Sibling | 3 | 3 | 3 | 3 | 12
    Parent | 2 | 6 | 1 | 3 | 12
    Other | 8 | 8 | 12 | 12 | 40
Primary Diagnosis of Veteran [Count of Participants; unit: Participants] — Primary life-limiting diagnosis of Veteran patient Population: Primary diagnosis of veteran only collected from patient half of dyad, which =143
  Participants
    Cancer: number analyzed (Participants) | 0 | 71 | 0 | 72 | 143
    Cancer |  | 43 |  | 52 | 95
    Congestive Heart Failure: number analyzed (Participants) | 0 | 71 | 0 | 72 | 143
    Congestive Heart Failure |  | 6 |  | 6 | 12
    Chronic obstructive pulmonary disease: number analyzed (Participants) | 0 | 71 | 0 | 72 | 143
    Chronic obstructive pulmonary disease |  | 12 |  | 5 | 17
    End Stage Renal Disease: number analyzed (Participants) | 0 | 71 | 0 | 72 | 143
    End Stage Renal Disease |  | 6 |  | 6 | 12
    Multiple Qualifying Disease: number analyzed (Participants) | 0 | 71 | 0 | 72 | 143
    Multiple Qualifying Disease |  | 4 |  | 3 | 7
Education [Count of Participants; unit: Participants]
  HS or less | 34 | 33 | 28 | 31 | 126
  Some College | 22 | 25 | 31 | 29 | 107
  College Degree | 12 | 6 | 5 | 6 | 29
  Graduate Work or Degree | 3 | 7 | 8 | 6 | 24
Finances [Count of Participants; unit: Participants] — Self-reported household finances by participant
  Participants
    Difficulty paying bills | 10 | 13 | 6 | 6 | 35
    Money to pay bills, cut back on things | 13 | 14 | 22 | 13 | 62
    Enough to pay bills, little extras | 26 | 22 | 23 | 30 | 101
    enough to pay bills and special things | 22 | 22 | 21 | 22 | 87
    Missing | 0 | 0 | 0 | 1 | 1
Employment [Count of Participants; unit: Participants] — Self-reported employment
  Participants
    Working Full or Part Time | 21 | 1 | 19 | 4 | 45
    Retired/Not Working | 43 | 38 | 42 | 40 | 163
    Disabled | 7 | 32 | 10 | 28 | 77
    Other | 0 | 0 | 1 | 0 | 1
Self-rated Quality of Health [Count of Participants; unit: Participants]
  Excellent | 0 | 0 | 1 | 0 | 1
  Very Good | 10 | 1 | 13 | 4 | 28
  Good | 16 | 11 | 14 | 8 | 49
  Fair | 9 | 14 | 9 | 14 | 46
  Poor | 0 | 9 | 0 | 12 | 21
  Missing | 36 | 36 | 35 | 34 | 141
Years of caregiving given or received [Mean (Standard Deviation); unit: years] — Self-reported years spent caregiving or years received caregiving
  years | 4.6 (5.6) | 5.2 (5.95) | 3.7 (4.06) | 3.4 (4.2) | 4.2 (5.04)
Number of Hours patient requires assistance [Mean (Standard Deviation); unit: hours] — Self-reported number of hours patient requires assistance
  hours | 2.4 (1.24) | 2.3 (1.34) | 2.3 (1.2) | 2.1 (1.25) | 2.3 (1.26)

OUTCOME MEASURES:

1. Primary Outcome: Caregiver Anxiety
Description: Profile of Moods States (POMS) anxiety sub-scale The anxiety sub-scale from the modified Brief Profile of Mood States (POMS),7110 a six-item measure of psychological distress. Individual items used a 5 point Likert scale (0-4). The sub-scale minimum score was 0 and maximum was 24 (more anxious ).
Time Frame: Measured at baseline, 5 weeks, and 8 weeks
Population: Comparing Caregiver anxiety levels between the Outlook and the Relaxation meditation arm. Differences in numbers analyzed versus group totals due to missing data.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Caregiver Outlook - Caregiver: Three facilitator-led preparation and completion sessions with the caregiver discussing life review, issues of forgiveness and heritage and legacy (Intervention).
- Relaxation Meditation - Caregiver: Three facilitator-led sessions of caregivers listening to a non-guided relaxation CD (Attention Control).
Arm/Group | Caregiver Outlook - Caregiver | Relaxation Meditation - Caregiver
Number analyzed (Participants) | 71 | 71
units on a scale
  Baseline | 6.9 (5.3) | 7.3 (4.6)
  5 week follow up: number analyzed (Participants) | 54 | 52
  5 week follow up | 5.9 (5.2) | 5.4 (4.9)
  8 week follow up: number analyzed (Participants) | 60 | 56
  8 week follow up | 5.8 (5.7) | 6.4 (5.1)
Statistical Analysis 1: Comparison: Caregiver Outlook - Caregiver vs Relaxation Meditation - Caregiver; Note- missing the first follow up at 5 weeks did not prohibit an individual from participating at the second follow up at 8 weeks; Test type: Superiority or Other; p < 0.511, Mixed Models Analysis — Between Outlook Intervention and Attention Control caregivers at 5 weeks; Mean Difference (Final Values) = 0.5376, 95% CI 2-sided [-1.0776 to 2.1528]
Statistical Analysis 2: Comparison: Caregiver Outlook - Caregiver vs Relaxation Meditation - Caregiver; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.6348, Mixed Models Analysis — Between Outlook Intervention and Attention Control caregivers at 8 weeks; Mean Difference (Final Values) = 0.4275, 95% CI 2-sided [-1.3505 to 2.2055]

2. Secondary Outcome: Spirituality
Description: Functional Assessment of Chronic Illness Therapy - Spiritual Well-Being (FACIT-SP) subscale. The 12-item measure assess spiritual well-being: faith, meaning, and purpose. Individual items use a 5 point likert scale (0-4). The scale minimum score is 0 (negative well being) and maximum is 48 (positive well being).
Time Frame: Measured at baseline, 5 weeks, and 8 weeks
Population: Comparing spiritual well being levels between the Outlook and the Relaxation meditation arms, Caregivers only.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Caregiver Outlook - Caregiver | Relaxation Meditation - Caregiver
Number analyzed (Participants) | 71 | 72
units on a scale
  Baseline | 35.4 (9.0) | 37.3 (7.2)
  5 week: number analyzed (Participants) | 54 | 52
  5 week | 36.1 (8.0) | 37.3 (7.0)
  8 week: number analyzed (Participants) | 60 | 55
  8 week | 37.3 (8.3) | 36.6 (7.6)
Statistical Analysis 1: Comparison: Caregiver Outlook - Caregiver vs Relaxation Meditation - Caregiver; Comparison at 5 weeks Note- missing the first follow up at 5 weeks did not prohibit an individual from participating at the second follow up at 8 weeks; Test type: Superiority or Other; p = 0.5225, Mixed Models Analysis; Mean Difference (Final Values) = 0.6836, 95% CI 2-sided [-1.4278 to 2.7950]
Statistical Analysis 2: Comparison: Caregiver Outlook - Caregiver vs Relaxation Meditation - Caregiver; Comparison at 8 weeks. Note-missing the first follow up at 5 weeks did not prohibit an individual from participating at the second follow up at 8 weeks; Test type: Superiority or Other; p = 0.1972, Mixed Models Analysis; Mean Difference (Final Values) = 1.2764, 95% CI 2-sided [-0.6728 to 3.2257]

3. Secondary Outcome: Depression
Description: Centers for Epidemiologic Study of Depression short form (CES-D) is a 10-item measure of depression. Items are rated on a 4 point Likert scale (0-3) with total scores ranging from 0 to 30. Higher scores indicate greater depressive symptoms
Time Frame: Measured at baseline, 5 weeks, and 8 weeks
Population: Primary and secondary results are comparing caregiver scores in the two arms, not patient arms.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Caregiver Outlook - Caregiver | Relaxation Meditation - Caregiver
Number analyzed (Participants) | 71 | 72
units on a scale
  Baseline | 8.2 (6.6) | 8.8 (5.5)
  5 weeks: number analyzed (Participants) | 54 | 52
  5 weeks | 8.7 (6.8) | 8.0 (6.4)
  7 weeks: number analyzed (Participants) | 59 | 56
  7 weeks | 8.3 (6.2) | 9.0 (6.4)
Statistical Analysis 1: Comparison: Caregiver Outlook - Caregiver vs Relaxation Meditation - Caregiver; Between Outlook Intervention caregivers and active control caregivers at 5 weeks Note- missing the first follow up at 5 weeks did not prohibit an individual from participating at the second follow up at 8 weeks; Test type: Superiority or Other; p < 0.3332, Mixed Models Analysis; Mean Difference (Final Values) = 0.9358, 95% CI 2-sided [-0.9726 to 2.8443]
Statistical Analysis 2: Comparison: Caregiver Outlook - Caregiver vs Relaxation Meditation - Caregiver; Between Outlook Intervention caregivers and active control caregivers at 8 weeks Note - Missing the first follow up at 5 weeks did not prohibit an individual from participating at the second follow up at 8 weeks; Test type: Superiority or Other; p = 0.3842, Mixed Models Analysis — Note-missing the first follow up at 5 weeks did not prohibit an individual from participating at the second follow up at 8 weeks; Mean Difference (Final Values) = 0.6929, 95% CI 2-sided [-0.8783 to 2.2642]

4. Secondary Outcome: Patient Days of VA Hospital Use
Description: The number of days that a patient used either the VA emergency department (ED) or was an inpatient at a VA hospital in the 6 months following randomization. Inclusion of non-VA utilization was made unpractical due to the long delay in filing for non VA reimbursement (up to 2 years). The original variable was Day AT home, defined to be 180 days minus the days in ED or inpatient hospital. This was changed to days of use due to distribution/modeling considerations.
Time Frame: In the 6 months after randomization
Measure: Mean (Standard Deviation); unit: Days in VA hospital or ER
Groups:
- Caregiver Outlook - Patient: Three facilitator-led preparation and completion sessions with the caregiver discussing life review, issues of forgiveness and heritage and legacy (Intervention).
- Relaxation Meditation - Patient: Three facilitator-led sessions of caregivers listening to a non-guided relaxation CD (Attention Control).
Arm/Group | Caregiver Outlook - Patient | Relaxation Meditation - Patient
Number analyzed (Participants) | 71 | 72
Days in VA hospital or ER | 4.4 (11.8) | 4.4 (9.6)
Statistical Analysis 1: Comparison: Caregiver Outlook - Patient vs Relaxation Meditation - Patient; Test type: Superiority or Other; p = 0.8748, Standard negative binomial with offset; expected change in difference in logs = 0.0593, 95% CI 2-sided [-0.6784 to 0.797] — The expected change in the difference of the logs of expected Days in VA inpatient care or ED

5. Secondary Outcome: Caregiver Burden
Description: Caregiver Reaction Assessment (CRA). The Caregiver Reaction Assessment is a 24-item multidimensional instrument designed to measure a caregiver's reactions to caregiving for family members with a variety of chronic illnesses. The esteem subscale has 7 items with a 5 level Likert scale: 1=Strongly Disagree to 5=Strongly Agree. The score is the average of the 7 items ranging from a low score of 1 associated with negative reactions and high score of 5 with positive reactions.
Time Frame: Measured at baseline, 5 weeks, and 8 weeks
Population: Comparing Caregiver reaction assessment scores between the Outlook Intervention and the Relaxation Meditation arm.Differences in numbers analyzed versus group totals due to missing data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Caregiver Outlook - Caregiver | Relaxation Meditation - Caregiver
Number analyzed (Participants) | 70 | 70
units on a scale
  Baseline | 4.2 (0.6) | 4.2 (0.6)
  5 week: number analyzed (Participants) | 53 | 52
  5 week | 4.2 (0.6) | 4.2 (0.6)
  8 week: number analyzed (Participants) | 57 | 56
  8 week | 4.2 (0.6) | 4.1 (0.6)
Statistical Analysis 1: Comparison: Caregiver Outlook - Caregiver vs Relaxation Meditation - Caregiver; Between Outlook Intervention caregivers and active control caregivers at 5 weeks. Note- missing the first follow up at 5 weeks did not prohibit an individual from participating at the second follow up at 8 weeks; Test type: Superiority or Other; p = 0.7687, Mixed Models Analysis — Between Caregiver Outlook - Caregiver and Relaxation Meditation - Caregiver at 5 weeks; Mean Difference (Final Values) = -0.01777, 95% CI 2-sided [-0.1372 to 0.1017]
Statistical Analysis 2: Comparison: Caregiver Outlook - Caregiver vs Relaxation Meditation - Caregiver; Between Outlook Intervention caregivers and active control caregivers at 8 weeks Note- missing the first follow up at 5 weeks did not prohibit an individual from participating at the second follow up at 8 weeks; Test type: Superiority or Other; p = 0.9863, Mixed Models Analysis — Between Caregiver Outlook - Caregiver and Relaxation Meditation - Caregiver at 8 weeks; Mean Difference (Final Values) = -0.00087, 95% CI 2-sided [-0.1003 to 0.09861]

6. Secondary Outcome: Caregiver Completion
Description: Quality of life at the End of Life (Family Edition) is a 17-item measure of quality of life at the end of life assessing five domains: life completion, relationship with health care providers, preparation for death, physical symptoms and affective social support. The 3-item Life Completion subscale uses a 5 point (0-4) Likert scale. The subscale ranges from 0 (poor) to 4 (better outcome).
Time Frame: Measured at baseline, 5 weeks, and 8 weeks
Population: Comparing life completion scores between the Outlook Intervention and the Relaxation meditation arm, caregivers only. Differences in numbers analyzed versus group totals due to missing data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Caregiver Outlook - Caregiver | Relaxation Meditation - Caregiver
Number analyzed (Participants) | 70 | 71
units on a scale
  Baseline | 2.7 (0.8) | 2.8 (0.8)
  5 Week: number analyzed (Participants) | 54 | 52
  5 Week | 2.5 (0.9) | 2.6 (0.9)
  8 Week: number analyzed (Participants) | 59 | 56
  8 Week | 2.5 (1.0) | 2.7 (0.8)
Statistical Analysis 1: Comparison: Caregiver Outlook - Caregiver vs Relaxation Meditation - Caregiver; At 5 weeks - Completion subscale; Test type: Superiority or Other; p = 0.9221, Mixed Models Analysis; Mean Difference (Final Values) = -0.01166, 95% CI 2-sided [-0.2475 to 0.2241]
Statistical Analysis 2: Comparison: Caregiver Outlook - Caregiver vs Relaxation Meditation - Caregiver; Comparison at 8 week time point Note- Missing first follow up at 5 weeks did not prohibit an individual from participating at the second follow up at 8 week; Test type: Superiority or Other; p = 0.3249, Mixed Models Analysis — Between Caregiver Outlook - Caregiver and Relaxation Meditation - Caregiver at 8 weeks; Mean Difference (Final Values) = -0.1154, 95% CI 2-sided [-0.3466 to 0.1158]

7. Secondary Outcome: Prolonged Grief - Number of Participants With Anticipatory Grief
Description: The Prolong Grief Disorder scale is a clinically-based diagnosis determination scale modified for this study. The components/requirements that were dropped were a) diagnosis should not be made until at least 6 months since death, and b) the disturbance is not better accounted for major depressive disorder, generalized anxiety disorder or post traumatic stress disorder. The outcome was a dichotomized variable with 1 indicating symptoms of prolonged grief are present and 0 indicating insufficient symptoms.
Time Frame: Measured at baseline, 5 weeks, and 8 weeks
Population: Number of participants indicating prolonged grief across the Outlook Intervention and the Relaxation meditation arm, caregivers only. Only six percent of the sample qualified as having prolonged grief, at baseline. Therefore there was not sufficient data for statistical modeling.
Measure: Number; unit: participants
Arm/Group | Caregiver Outlook - Caregiver | Relaxation Meditation - Caregiver
Number analyzed (Participants) | 71 | 72
participants
  Baseline | 6 | 2
  5 week: number analyzed (Participants) | 54 | 52
  5 week | 2 | 3
  8 week: number analyzed (Participants) | 59 | 56
  8 week | 2 | 2

8. Secondary Outcome: Caregiver Preparation
Description: Quality of life at the End of Life (Family Edition) is a 17-item measure of quality of life at the end of life assessing five domains: life completion, relationship with health care providers, preparation for death, physical symptoms and affective social support. The 5-item preparation subscale uses a 5 point (0-4) Likert scale. The subscale ranges from 0 (poor) to 4 (better outcome).
Time Frame: Measured at baseline, 5 weeks, and 8 weeks
Population: Comparing preparation scores between the Outlook Intervention and the Relaxation meditation arm, caregivers only. Two scale items were inadvertently left out initially. Items were added back in when omission was noted. However, the large number of missing makes analysis inappropriate.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Caregiver Outlook - Caregiver | Relaxation Meditation - Caregiver
Number analyzed (Participants) | 36 | 37
units on a scale
  Baseline: number analyzed (Participants) | 33 | 37
  Baseline | 2.7 (0.7) | 2.4 (0.8)
  5 Week: number analyzed (Participants) | 34 | 28
  5 Week | 2.4 (0.8) | 2.7 (0.7)
  8 Week: number analyzed (Participants) | 36 | 30
  8 Week | 2.6 (0.8) | 2.6 (0.8)

ADVERSE EVENTS:
Time Frame: During time of study participation, 8 weeks per participant. Adverse events were collected both systematically, by asking of events at each time point, and non-systematically.
Groups:
- Caregiver Outlook - Caregiver: Intervention: Three facilitator-led sessions with the caregiver discussing life review, issues of forgiveness and heritage and legacy.
- Caregiver Outlook - Patient: Patients of the caregivers in the Outlook Intervention arm.
- Relaxation Meditation - Patient: Patients of the caregivers in the Attention Control arm.
Arm/Group | Caregiver Outlook - Caregiver | Caregiver Outlook - Patient | Relaxation Meditation - Caregiver | Relaxation Meditation - Patient
Serious Adverse Events (participants affected / at risk) | 0/71 | 13/71 | 0/72 | 11/72
Other Adverse Events (participants affected / at risk) | 4/71 | 7/71 | 4/72 | 11/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Caregiver Outlook - Caregiver (N=71) | Caregiver Outlook - Patient (N=71) | Relaxation Meditation - Caregiver (N=72) | Relaxation Meditation - Patient (N=72)
Cardiac (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Gastro-Intestinal (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (6) | 0 (0) | 3 (5)
Renal (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Respiratory (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Surgery (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neoplasm-death (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 4 (4) | 0 (0) | 3 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Caregiver Outlook - Caregiver (N=71) | Caregiver Outlook - Patient (N=71) | Relaxation Meditation - Caregiver (N=72) | Relaxation Meditation - Patient (N=72)
Infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 7 (7)
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 5 (5) | 0 (0) | 3 (5)
Psychiatric (Psychiatric disorders) | 4 (6) | 0 (0) | 4 (5) | 0 (0)
Vascular/blood (Vascular disorders) | 0 (0) | 5 (6) | 0 (0) | 1 (1)
Multiple/general (General disorders) | 0 (0) | 4 (4) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes